CLINICAL TRIAL: NCT06714630
Title: Improving Radiotherapy in PROState Cancer Using EleCtronic Population-based healthCAre Data: The PROSECCA Study, Answering New Questions in Prostate Cancer
Brief Title: The PROSECCA Study, Answering New Questions in Prostate Cancer
Acronym: PROSECCA
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); NHS Grampian (Other Government); NHS Highland (Other); NHS Tayside (Other Government); University of Glasgow (Other); University of Lyon (Other); NHS Lothian (Other Government); NHS Research Scotland (Other); Public Health Scotland (Unknown); Prostate Cancer UK (Other); Movember Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0221
Record Dates: First submitted 2024-08-13; First posted 2024-12-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Artificial Intelligence; Radiotherapy reactions; clinical decisions; predict outcomes; Patient individualised response; Machine Learning; AI; Personalized Radiotherapy; Radiotherapy Adaptation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nearly half of all cancer patients receive radiotherapy as part of their treatment and although it is effective at destroying cancerous lesions deep within the body, this comes at the cost of damaging healthy, or normal, tissues. With 50% of cancer patients surviving for 10 years or more, these patients can be left with life-changing side effects from their radiotherapy. It is clear that more must be done to limit damage to normal healthy tissue without compromising annihilation of the tumour and curing patients. The key to this is personalising an individual's radiotherapy treatment, in other words rather than assuming that all tumours respond similarly to radiotherapy, the treatment is optimised for an individual. To date, approaches to do this have been restricted to small numbers of carefully selected patients, are inordinately expensive, and not suitable for rolling out into everyday practice across the NHS. There is however another way, namely using Artificial Intelligence (AI) combined with an individual's healthcare record. By linking together large numbers of healthcare records at a national level, combined with the power of AI, the PROSECCA project will transform radiotherapy and cancer care.

DETAILED DESCRIPTION:
As an example of how this technology is beginning to emerge, proof of concept data from the team has shown that using AI it is possible to identify patients at increased risk of damage from radiotherapy long before they receive any radiation as part of their treatment. However, to move these AI-based approaches from the research domain into the clinic requires significant effort, which is the aim of PROSECCA study.

The project will use AI to analyse healthcare records from up to 15,000 prostate cancer patients who underwent radiotherapy in Scotland. Through linkage of data obtained specifically for radiotherapy and data held within each patient's unique healthcare history it will be possible to establish new relationships between a patient's medical history and how well a patient responds to radiotherapy. By establishing what factors or information in a patient's complex healthcare record indicate that an individual may have a poor response to treatment, or an increased risk of side effects from radiation, it will be possible to identify these patients earlier than is currently possible and adapt treatment accordingly. Furthermore, identifying these important factors would improve radiotherapy treatment for prostate cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* External beam radiotherapy delivered by a linear accelerator
* Prostate Specific Antigen (PSA) recorded at regular intervals after radiotherapy
* Minimum of 10 year survival post-radiotherapy
* Diagnostic Computerised Tomography (CT) acquired
* Radiotherapy planning CT acquired
* Radiotherapy treatment planning data available
* Corresponding healthcare data available to infer toxicity events (ref previous work by Lemanska et al)

Exclusion Criteria:

* Incomplete course of radiotherapy
* No PSA data
* No follow-up corresponding healthcare data available
* No imaging data available

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study requires no new data to be acquired relying solely on data collected on previously treated prostate cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
PSA relapse free survival | Plus/minus 10 years from date of radiotherapy treatment
  PSA relapse free survival will be measured from the date of treatment. This information will be obtained from historical patient records.
  The expected number of events in this category was calculated using the following approach.
  5 year endpoint, 10% event rate based on Conventional or hypofractionated high dose intensity modulated radiotherapy for prostate cancer (CHHIP) trial Data up to 2015 resulting in sample size of 11,250 (75% of 15,000) Total Events = 1125
Overall Survival | Plus/minus 10 years from date of radiotherapy treatment
  Overall survival will be measured from the date of treatment. This information will be obtained from historical patient records.
  The expected number of events in this category was calculated using the following approach.
  10 year endpoint, 29% event rate based on RT01 radiotherapy trial Data up to 2010 resulting in sample size of 7,500 (50% of 15,000) Total Events = 2175
Radiotherapy Toxicity | Plus/minus 10 years from date of radiotherapy treatment
  Radiotherapy Toxicity was estimated based on the cohort toxicity reported in the CHHIP trial. The same estimates were applied to this cohort with the expected number of events as follows.
  Note that a higher attrition rate is expected for this endpoint, 60% of 15,000=10,000 5 year endpoint, 12% event rate for Grade 2+ toxicity based on CHHIP trial Total Events = 900

CONTACTS AND LOCATIONS:
Overall Officials: Bill Nailon, Principal Investigator — University of Edinburgh; Duncan McLaren, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Derived] Nailon WH, Noble DJ, Harrison E, Yang Z, Elliot S, MacNair A, Beckett G, Hallam A, Sheikh A, Mills N, Halliday R, Morrison D, Chalmers A, Cameron D, Gourley C, Hall P, Lilley C, Carruthers LJ, Trainer M, Burns D, Dee F, Andiappa S, Lonsdale A, Couper M, Farnan K, McLellan J, Miller A, Ogg J, Moses J, Colligan S, MacDonald G, McPhail N, Niblock P, MacLeod N, Davies ME, Laurenson DI, Hopgood JR, Boyle D, Paterson C, Grose D, Phillips I, Harrow S, Berger T, Shelley LEA, Sanders I, Henderson S, Duffton A, Mitchell J, Rutherford A, McLaren DB. Protocol for the PROSECCA study: a new approach for predicting radiotherapy outcome using artificial intelligence and electronic population-based healthcare data. BMJ Open. 2026 Feb 2;16(2):e104408. doi: 10.1136/bmjopen-2025-104408. PMID 41628931